CLINICAL TRIAL: NCT07337291
Title: Double Versus Single Plastic Stents for Non-Retrievable Biliary Stones in Cirrhotic Patients
Brief Title: Double Stent for Biliary Stones in Cirrhotic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01282612295; 00787 (Registry Identifier: The Institution Review Board of National Liver Institute, Menoufia University, Egypt)
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Liver Circulation; Choledocholithiasis; Stent
Keywords: ERCP; Biliary Stent; Double Stent; Liver Cirrhosis; Non-Retrievable Stones; High-Risk Patients
MeSH Terms: conditions — Choledocholithiasis; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single 10 Fr Plastic Stent (Experimental): Placement of a single 10 French (Fr), 10 cm plastic biliary stent.
  Interventions: Device: Single 10 Fr Plastic Biliary Stent
- Double 10 Fr Plastic Stents (Experimental): Placement of two 10 French (Fr), 10 cm plastic biliary stents side-by-side.
  Interventions: Device: Two 10 Fr Plastic Biliary Stent
- Single 11.5 Fr Plastic Stent (Experimental): Placement of a single 11.5 French (Fr), 10 cm plastic biliary stent.
  Interventions: Device: Single 11.5 Fr Plastic Biliary Stent
- Single 10 Fr Pigtail Stent (Experimental): Placement of a single 10 French (Fr), 10 cm pigtail plastic biliary stent.
  Interventions: Device: Single 10 Fr Pigtail Stent

INTERVENTIONS:
Device: Single 10 Fr Plastic Biliary Stent — Single 10 Fr, 10 cm plastic stent placed endoscopically.
  Arms: Single 10 Fr Plastic Stent
Device: Two 10 Fr Plastic Biliary Stent — Two 10 Fr, 10 cm plastic stents placed endoscopically.
  Arms: Double 10 Fr Plastic Stents
Device: Single 11.5 Fr Plastic Biliary Stent — Single 11.5 Fr, 10 cm plastic stent placed endoscopically.
  Arms: Single 11.5 Fr Plastic Stent
Device: Single 10 Fr Pigtail Stent — Single 10 Fr, 10 cm pigtail plastic stent placed endoscopically.
  Arms: Single 10 Fr Pigtail Stent

SUMMARY:
This prospective, single-center, interventional study enrolled 400 cirrhotic patients with large or complex common bile duct (CBD) stones that could not be removed during an initial Endoscopic Retrograde Cholangiopancreatography (ERCP). The study compared four different plastic biliary stenting strategies (single 10 Fr, double 10 Fr, single 11.5 Fr, and single 10 Fr pigtail stents) to determine the optimal approach for facilitating successful stone clearance in a subsequent ERCP and minimizing complications in this high-risk patient population.

DETAILED DESCRIPTION:
Background and Rationale: The primary treatment for choledocholithiasis is Endoscopic Retrograde Cholangiopancreatography (ERCP) with sphincterotomy. However, complete stone clearance fails in 10-15% of cases involving complex choledochal stones (e.g., larger than 15 mm and/or more than 3 stones), often necessitating recurrent ERCP procedures. This challenge is compounded in high-risk patients, such as the elderly or those with substantial comorbidities, who cannot tolerate prolonged procedures. Failure to extract stones can also be attributed to anatomical factors like complex stones, periampullary diverticula, or ductal anomalies. While alternative methods like ESWL or lithotripsy exist, they are not universally available. Temporary plastic biliary stent placement is a safe and effective alternative, providing biliary drainage and acting as a bridge to subsequent stone removal. Short-term stenting can reduce stone size and improve the success rate of later extraction.

The aim of this work is to evaluate the role and efficiency of different types or different numbers of plastic stent application in the treatment of non-retrievable large biliary stones in liver cirrhosis.

Study Design and Setting: This is a prospective, single-center, interventional study conducted at the National Liver Institute, Menoufia University, Egypt, between January 2022 and January 2025. The study was authorized by the Institutional Ethics Committee (Approval No.: 00787/2025). A total of 400 cirrhotic patients with calculous biliary obstruction were included. Study Population and Eligibility: Participants were adults with established liver cirrhosis classified as high-risk due to moderate to severe liver disease and/or substantial comorbidities, who could not safely tolerate extended endoscopic or surgical intervention. They all presented with large or complex Common Bile Duct (CBD) stones that could not be removed during the initial ERCP. All enrolled subjects were clinically stable and provided signed informed consent. Exclusion criteria included non-cirrhotic patients, non-calculous causes of biliary obstruction (e.g., portal biliopathy, malignant obstruction), acute suppurative cholangitis, ERCP contraindications, or inability to complete the scheduled 12-month follow-up.

Interventions and Study Groups: Enrolled individuals were allocated into four parallel groups based on the type and size of the plastic biliary stent used during ERCP: Group 1 (Single plastic stent, 10 cm × 10 Fr), Group 2 (Double plastic stents, each 10 cm × 10 Fr), Group 3 (Single plastic stent, 10 cm × 11.5 Fr), and Group 4 (Single pigtail stent, 10 cm × 10 Fr). ERCP Procedure: All ERCPs were performed by expert hepatobiliary endoscopists under general anesthesia using a standard side-viewing duodenoscope. Following selective CBD cannulation, stone extraction was attempted. When complete clearance was not achievable, the appropriate plastic stent(s) were placed over a guidewire, with or without a previous sphincterotomy. Prolonged procedures, advanced lithotripsy techniques, and chemical stone dissolution were deliberately avoided due to the high-risk nature of the study population. Data Collection and Follow-up: Thorough clinical and demographic data were systematically documented. Baseline laboratory investigations included renal function tests, CBC, CRP, pancreatic enzymes, and a full liver biochemical profile. Imaging (ultrasonography and MRCP) was used to characterize stone size, number, and biliary anatomy. Patients were observed for a minimum of 24 hours post-procedure. Follow-up assessments were scheduled at 1 month and subsequently at 3-6 month intervals or on demand. The total monitoring period was 12 months, with the final assessment completed by January 2026. Follow-up involved clinical assessment, laboratory tests, and abdominal radiographs to assess biliary drainage and stent patency. Patients with signs of stent malfunction underwent repeat ERCP.

Outcome Measures: The main outcomes were stent patency and successful stone clearance at the second ERCP. Secondary objectives included reduction in stone size, all-cause mortality throughout the follow-up period, and procedure-related complications (stent migration, cholangitis, post-ERCP pancreatitis, and hemorrhage).

Statistical Analysis: Statistical analysis will be performed using IBM SPSS Statistics (version 22). Comparisons among groups will be completed using the chi-square (χ²) test or Monte Carlo correction for categorical variables, one-way ANOVA for normally distributed continuous variables, and the Kruskal-Wallis test for non-normally distributed variables. A p-value ≤ 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with established liver cirrhosis.
2. Presence of large or complex common bile duct (CBD) stones that were non-retrievable during the initial ERCP.
3. Classified as high-risk due to moderate to severe liver disease and/or substantial comorbidities, making them unable to safely tolerate extended endoscopic procedures or surgical intervention.
4. Clinically stable and capable of undergoing the scheduled diagnostic and therapeutic procedures.
5. Provided signed informed consent before enrollment.

Exclusion Criteria:

1. Non-cirrhotic patients.
2. Patients with non-calculous causes of biliary obstruction (e.g., portal biliopathy, benign biliary strictures, or malignant biliary obstruction).
3. Acute suppurative cholangitis.
4. Contraindications to ERCP.
5. Inability to complete the scheduled 12-month follow-up time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Stent Patency | 6 months
  Time from stent placement until clinical or biochemical evidence of stent occlusion (e.g., cholangitis, elevated liver enzymes, or imaging findings).
Successful Stone Clearance in Second ERCP | 6 months
  The proportion of patients in each group achieving complete clearance of common bile duct stones during the second, planned ERCP session.

SECONDARY OUTCOMES:
Incidence of Procedure-Related Complications | From stenting until 30 days after the second ERCP.
  Incidence of adverse events, including stent migration, cholangitis, post-ERCP pancreatitis, and hemorrhage.
Reduction in Stone Size | 6 months
  Mean reduction in the largest stone diameter, measured by cholangiography or MRCP, between initial stenting and the second ERCP.
All-Cause Mortality | 12 months
  The number of deaths from any cause during the study follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- National Liver Institute, Menoufia University, Egypt., Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee TH, Han JH, Kim HJ, Park SM, Park SH, Kim SJ. Is the addition of choleretic agents in multiple double-pigtail biliary stents effective for difficult common bile duct stones in elderly patients? A prospective, multicenter study. Gastrointest Endosc. 2011 Jul;74(1):96-102. doi: 10.1016/j.gie.2011.03.005. Epub 2011 Apr 30. PMID 21531412
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Kato N, Kamijima T, Graham DY, Tanaka N. Biliary stenting in the management of large or multiple common bile duct stones. Gastrointest Endosc. 2010 Jun;71(7):1200-1203.e2. doi: 10.1016/j.gie.2009.12.055. Epub 2010 Apr 18. PMID 20400079
- [Background] Binmoeller KF, Schafer TW. Endoscopic management of bile duct stones. J Clin Gastroenterol. 2001 Feb;32(2):106-18. doi: 10.1097/00004836-200102000-00004. PMID 11205644